CLINICAL TRIAL: NCT06280846
Title: High-intensity Versus Low-intensity Laser Acupuncture in Chronic, Non-specific Low Back Pain: a Double-blinded, Randomized Controlled Trial
Brief Title: High-intensity Versus Low-intensity Laser Acupuncture in Chronic, Non-specific Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: King Khalid University (Other)
Responsible Party: Principal Investigator, Doaa Ayoub Elimy Mohammed, Lecturer of physical therapy for basic science department., faculty of physical Therapy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/004878
Record Dates: First submitted 2024-02-16; First posted 2024-02-28 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Chronic Nonspecific Low-back Pain
Keywords: low back pain; high-intensity laser acupuncture; Low-intensity laser acupuncture; peak torque; fatigue; functional disability
MeSH Terms: conditions — Low Back Pain; Fatigue | interventions — Low-Level Light Therapy

STUDY DESIGN:
Intervention Model Description: high-intensity laser acupuncture, low-intensity laser acupuncture and exercise therapy program
Who Masked: Participant, Outcomes Assessor
Masking Description: random generator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental high-intensity laser acupuncture and an exercise therapy program. (Experimental): The patients will receive high-intensity laser acupuncture and an exercise therapy program.three times a week for four weeks.
  Interventions: Device: high-intensity laser acupuncture and Exercise therapy program
- Experimental low-intensity laser acupuncture and an exercise therapy program. (Experimental): The patients will receive low-intensity laser acupuncture and an exercise therapy program.three times a week for four weeks.
  Interventions: Device: low-intensity laser acupuncture and Exercise therapy program
- sham laser acupuncture and an exercise therapy program. (Sham Comparator): The patients will receive a sham laser acupuncture and an exercise therapy program three times a week for four weeks.
  Interventions: Device: Sham laser acupuncture

INTERVENTIONS:
Device: high-intensity laser acupuncture and Exercise therapy program — The patients will receive high-intensity lasers and the treatment will be performed at 15 acupuncture points: unilateral GV3, GV4, and GV5, and bilateral BL 20, BL23, BL24, BL25, BL40 and GB30.
  Exercise therapy program: The patients will perform an exercise therapy program in the form of:
  - strengthening exercises for abdominal and back muscles, - lumbar stabilization exercises. - stretching exercises
  Other Names: high-power laser acupuncture
  Arms: Experimental high-intensity laser acupuncture and an exercise therapy program.
Device: low-intensity laser acupuncture and Exercise therapy program — The patients will receive low-intensity lasers and the treatment will be performed at 15 acupuncture points: unilateral GV3, GV4, and GV5, and bilateral BL 20, BL23, BL24, BL25, BL40 and GB30.
  Exercise therapy program: The patients will perform an exercise therapy program in the form of:
  - strengthening exercises for abdominal and back muscles, - lumbar stabilization exercises. - stretching exercises
  Other Names: low power laser
  Arms: Experimental low-intensity laser acupuncture and an exercise therapy program.
Device: Sham laser acupuncture — Sham laser acupuncture and exercise therapy program. The patients will receive a sham laser.acupuncture and an exercise therapy program in the form of: - strengthening exercises for abdominal and back muscles, - lumbar stabilization exercises. - stretching exercises
  Arms: sham laser acupuncture and an exercise therapy program.

SUMMARY:
The purpose of this study is to investigate the efficacy of high-intensity laser acupuncture versus low intensity laser acupuncture on peak torque of trunk extensors, fatigue of trunk extensors, back pain, ROM and function in patients with chronic nonspecific low back pain (CNLBP).

DETAILED DESCRIPTION:
Chronic nonspecific low back pain is a type of persistent back pain that affects people of all ages and contributes to the global disease burden (CNLBP). The major objective of treatment is to lessen pain and its aftereffects. One noninvasive, targeted light therapy for treating musculoskeletal disorders is low-intensity laser therapy (LLLT). It has analgesic, anti-inflammatory, muscle-relaxant, and tissue-repair properties. Additionally, LILT has been demonstrated to relieve generalized lower back pain. Another light therapy that is painless and noninvasive, high-intensity laser therapy (HILT), stimulates tissue while delivering analgesic, anti-inflammatory, and anti-edematous benefits. It has been demonstrated that acupuncture, a popular complementary therapy, can relieve musculoskeletal pain and increase muscle strength.To date, however, there has been limited investigation into the effects of high- versus low-intensity laser acupuncture on CNLBP. Thus, the current study will be conducted to explore the efficacy of HILT versus LILL on peak torque of trunk extensors, fatigue of trunk extensors, back pain, ROM and functional disability in patients with chronic, nonspecific low back pain.

ELIGIBILITY:
Inclusion Criteria:

1. The patients had CNSLBP with age from 20 to 40 years from both genders.
2. Patients will be referred from an orthopedist with diagnosis of chronic low back pain without underlying pathological causes.
3. The patients with chronic nonspecific low back pain more than 3months. Minimum pain intensity of 30 mm on the visual analogue scale (VAS) for pain, which ranges from 0 to 100 mm.
4. Patients with normal BMI ranges between 18.5:24.9 kg/m2.
5. The study populations must be willing to participate in the study

Exclusion Criteria:

1. Neurological, infectious diseases and systemic illness such as rheumatologic diseases,systemic lupus erythematosus, diabetes mellitus type I or II.
2. Psychiatric/mental deficit.
3. Patients who had a previous surgical history (within 6 months) will also excluded.
4. participation in other treatment within the previous 3 month.
5. Pregnancy.
6. History of spinal fracture, tumor, osteoporosis

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2024-03-15 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
peak torque | up to four weeks
  Isokinetic dynamometer will be used for measuring peak torque of back extensors.
peak torque | follow up after 1 month
  Isokinetic dynamometer will be used for measuring peak torque of back extensors.
Fatigue | up to four weeks
  Isokinetic dynamometer will be used for measuring fatigue of back extensors.
Fatigue | follow up after 1 month
  Isokinetic dynamometer will be used for measuring fatigue of back extensors.

SECONDARY OUTCOMES:
Pain Intensity | up to four weeks
  Visual Analogue Scale (VAS) will be used by the patient to mark his/her level of pain between 0 to100 milliliters line.
  Zero usually represents 'no pain at all' whereas the upper limit represents 'the worst pain ever possible'.
Pain Intensity | follow up after 1 month
  Visual Analogue Scale (VAS) will be used by the patient to mark his/her level of pain between 0 to100 milliliters line.
  Zero usually represents 'no pain at all' whereas the upper limit represents 'the worst pain ever possible'.
lumbar flexion ROM assessment | up to four weeks
  Modified Schober test will be used to assess ROM of lumbar flexion.
lumbar flexion ROM assessment | follow up after 1 month
  Modified Schober test will be used to assess ROM of lumbar flexion.
Disability | up to four weeks
  Arabic version of Oswestry Disability Index (ODI) will be used for assessment of functional disability
Disability | follow up after 1 month
  Arabic version of Oswestry Disability Index (ODI) will be used for assessment of functional disability

CONTACTS AND LOCATIONS:
Locations (1):
- Doaa Ayoub Elimy, Giza, Egypt